CLINICAL TRIAL: NCT01449370
Title: A Phase I, Dose Escalation Study of MLN1117 in Subjects With Advanced Solid Malignancies Followed by Expansion in Subjects With Measurable Disease
Brief Title: Dose Escalation Study of TAK-117 (MLN1117) in Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INK1117-001
Record Dates: First submitted 2011-08-11; First posted 2011-10-10 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Solid Tumors
Keywords: INK1117; PIK3CA; KINASE; TUMOR; CANCER; Locally advanced or metastatic solid tumors; not eligible for standard of care therapy
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Neoplasms | interventions — serabelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): TAK-117 administered once a day orally
  Interventions: Drug: TAK-117
- Arm B (Experimental): TAK-117 administered orally intermittently, once every other day (Monday, Wednesday, and Friday) each week
  Interventions: Drug: TAK-117
- Arm C (Experimental): TAK-117 administered orally intermittently, once a day for 3 consecutive days (Monday, Tuesday, and Wednesday) each week
  Interventions: Drug: TAK-117

INTERVENTIONS:
Drug: TAK-117 — oral administration of TAK-117, daily and intermittent schedules.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and/or optimal biologic dose(OBD), safety and tolerability, dose-limiting toxicity (DLT) of TAK-117 when administered orally in subjects with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have had their PIK3CA gene mutation status assessed prior to enrolling into the study
* Subjects must have documented disease progression prior to enrolling into the study
* locally advanced or metastatic solid tumors with the exception of primary brain tumor, and have failed or are not eligible for standard of care therapy.
* Age greater than or equal to (>=) 18 years, including males and females;
* Eastern cooperative oncology group (ECOG) performance status (PS) 0-1;
* Adequate organ function;
* Male subjects must be surgically sterile or must agree to use physician-approved contraception during the study and for 30 days following the last study drug administration;
* Ability to swallow oral medications;
* Ability to understand and willingness to sign informed consent prior to initiation of any study procedures;
* For women of child-bearing potential, negative serum pregnancy test within 14 days prior to the first study drug administration and use of physician-approved method of birth control from 30 days prior to the first study drug administration to 30 days following the last study drug administration

Exclusion Criteria:

* Diagnosis of primary brain tumor; untreated brain metastasis or history of leptomeningeal disease or spinal cord compression;
* Received prior cancer or other investigational therapy within 2 weeks prior to the first administration of study drug;
* Have received a systemic corticosteroid within one week prior to the first administration of study drug;
* Clinically significant cardiac disease;
* Myocardial infarction or unstable angina within 6 months prior to the first administration of study drug;
* Malabsorption ;
* Poorly controlled diabetes mellitus;
* Pregnancy (positive serum or urine pregnancy test) or breast feeding;
* Untreated brain metastasis or history of leptomeningeal disease or spinal cord compression;
* Failed to recover from the reversible effects of prior anticancer therapies;
* Have received a selective phosphoinositide-3-kinase alpha isoform (PI3K-alpha) inhibitor
* Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system (CNS) disease, active infection, or any other condition that could compromise the subject's participation in the study
* Known human immunodeficiency virus (HIV) infection
* Have a secondary malignancy within the last 3 years prior to first dose of study drug, excluding treated non-melanoma skin cancer, carcinoma in situ, or locally-treated prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-10; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (5):
- United States (3):
  - Boston, Massachusetts
  - Detroit, Michigan
  - Dallas, Texas
- Barcelona, Spain
- Sutton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in England, Spain and the United States from 06 October 2011 to 15 January 2016.
Pre-assignment Details: Participants with advanced solid tumors were enrolled in dose escalation phase to receive TAK-117(MLN1117) in 1 of 4 treatment regimen.Study originally used clinical trial material(CTM) in Process A and new CTM in Process B. Due to limited single-agent TAK-117 activity in dose escalation phase,Study was terminated before start of planned expansion.
Groups:
- Process A: TAK-117 100 Milligram (mg), Once Daily (QD): TAK-117 100 mg, capsules (Process A), orally, QD up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process A: TAK-117 150 mg, QD: TAK-117 150 mg, capsules (Process A), orally, QD up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process A: TAK-117 200 mg, QD: TAK-117 200 mg, capsules (Process A), orally, QD up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process A: TAK-117 300 mg, QD: TAK-117 300 mg, capsules (Process A), orally, QD up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process A: TAK-117 200 mg, MWF QW: TAK-117 200 mg, capsules (Process A), orally, once every other day on Monday, Wednesday, and Friday each week (MWF QW) up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 300 mg, MWF QW: TAK-117 300 mg, capsules (Process A), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 400 mg, MWF QW: TAK-117 400 mg, capsules (Process A), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 600 mg, MWF QW: TAK-117 600 mg, capsules (Process A), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 900 mg, MWF QW: TAK-117 900 mg, capsules (Process A), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 1200 mg, MWF QW: TAK-117 1200 mg, capsules (Process A), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 200 mg, MTW QW: TAK-117 200 mg, capsules (Process A), orally, QD for 3 consecutive days, on Monday, Tuesday, and Wednesday each week (MTW QW) up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 400 mg, MTW QW: TAK-117 400 mg, capsules (Process A), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 600 mg, MTW QW: TAK-117 600 mg, capsules (Process A), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process A: TAK-117 900 mg, MTW QW: TAK-117 900 mg, capsules (Process A), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days.
- Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW: TAK-117 600 mg, capsules (Process B), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 900 mg FM MWF QW: TAK-117 900 mg, capsules (Process B), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 1200 mg FM MWF QW: TAK-117 1200 mg, capsules (Process B), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 600 mg FM MTW QW: TAK-117 600 mg, capsules (Process B), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 900 mg FM MTW QW: TAK-117 900 mg, capsules (Process B), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 1200 mg FM MTW QW: TAK-117 1200 mg, capsules (Process B), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 1500 mg FM MTW QW: TAK-117 1500 mg, capsules (Process B), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW: TAK-117 300 mg, capsules (Process B), orally, BID every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 400 mg FM BID MWF QW: TAK-117 400 mg, capsules (Process B), orally, intermittently, BID every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 500 mg FM BID MWF QW: TAK-117 500 mg, capsules (Process B), orally, intermittently, BID every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 600 mg FM BID MWF QW: TAK-117 600 mg, capsules (Process B), orally, intermittently, BID every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycles were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
Period: Overall Study
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Started | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
Not completed — Disease Progression | 5 | 4 | 8 | 3 | 3 | 3 | 3 | 2 | 9 | 1 | 3 | 3 | 2 | 8 | 3 | 1 | 4 | 3 | 1 | 2 | 5 | 2 | 3 | 7 | 3
Not completed — Adverse Event | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3
Not completed — Participant Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Medication Prohibited by Protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The all subjects as treated (ASaT) population included all enrolled participants who received at least 1 dose of TAK-117.
Groups:
- Total: Total of all reporting groups
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW | Total
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.79) | 59.0 (10.88) | 59.3 (9.05) | 45.3 (7.27) | 56.3 (17.67) | 52.7 (14.01) | 54.3 (12.58) | 65.0 (13.11) | 56.4 (13.28) | 53.3 (19.40) | 64.7 (18.58) | 50.0 (11.53) | 55.0 (9.54) | 57.4 (10.88) | 65.7 (12.86) | 62.7 (16.17) | 61.0 (11.89) | 52.7 (19.76) | 53.7 (1.53) | 66.7 (2.52) | 61.3 (13.68) | 72.5 (4.65) | 60.3 (11.81) | 66.0 (8.71) | 59.5 (10.39) | 59.4 (11.89)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 3 | 2 | 2 | 2 | 3 | 9 | 3 | 1 | 1 | 3 | 7 | 1 | 1 | 5 | 1 | 2 | 2 | 4 | 4 | 4 | 5 | 6 | 84
  Male | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 2 | 2 | 0 | 4 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 5 | 2 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 6 | 6 | 4 | 3 | 3 | 2 | 3 | 11 | 3 | 3 | 2 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 9 | 7 | 117
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 6 | 8 | 3 | 3 | 2 | 1 | 3 | 12 | 3 | 3 | 1 | 3 | 11 | 2 | 2 | 7 | 3 | 3 | 3 | 6 | 3 | 3 | 10 | 8 | 115
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Female Child Bearing Potential [Number; unit: participants]
  Females of Child-bearing Potential | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 7
  Post-menopausal | 4 | 3 | 3 | 0 | 1 | 1 | 1 | 1 | 4 | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 4 | 1 | 2 | 1 | 4 | 4 | 3 | 3 | 4 | 51
  Sterilized Females | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 2 | 4 | 1 | 1 | 0 | 1 | 5 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 26
  Males (Excluded from this analysis) | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 2 | 2 | 0 | 4 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 5 | 2 | 41
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Height data was available only for 119 participants as follow: n=5,6,8,2,3,2,3,3,12,3,3,3,3,11,3,3,7,3,3,3,6,4,4,9,7.
  centimeter (cm) | 161.70 (10.758) | 164.29 (7.241) | 165.25 (9.403) | 164.15 (5.837) | 164.19 (5.195) | 161.81 (5.222) | 165.17 (7.848) | 163.49 (6.883) | 163.08 (12.871) | 158.76 (9.161) | 168.76 (2.043) | 173.43 (6.072) | 164.67 (3.055) | 167.46 (10.274) | 170.22 (1.683) | 168.93 (16.176) | 168.32 (4.243) | 169.83 (13.829) | 169.52 (8.713) | 168.11 (6.887) | 165.97 (6.472) | 159.00 (3.939) | 157.05 (3.316) | 168.79 (13.186) | 164.87 (9.638) | 165.49 (9.098)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Weight data was available only for 123 participants as follow: n=5,6,8,4,3,2,3,3,12,3,3,3,3,11,3,3,7,3,3,3,6,4,4,10,8.
  kilogram (kg) | 62.18 (6.403) | 71.15 (21.862) | 73.48 (9.159) | 67.65 (24.513) | 72.48 (17.665) | 61.54 (2.487) | 57.73 (0.462) | 63.41 (3.880) | 69.14 (15.486) | 65.03 (15.137) | 70.76 (16.458) | 83.39 (28.852) | 60.60 (9.016) | 73.78 (12.955) | 72.26 (11.235) | 75.22 (12.679) | 79.84 (16.648) | 81.07 (25.417) | 82.72 (17.982) | 62.61 (15.706) | 64.59 (16.477) | 73.65 (16.747) | 65.37 (11.853) | 70.51 (15.263) | 65.11 (9.599) | 70.17 (14.958)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] — BSA data was available only for 119 participants as follow: n=5,6,8,2,3,2,3,3,12,3,3,3,3,11,3,3,7,3,3,3,6,4,4,9,7.
  square meter (m^2) | 1.67 (0.108) | 1.78 (0.266) | 1.83 (0.152) | 1.85 (0.500) | 1.81 (0.241) | 1.66 (0.060) | 1.63 (0.041) | 1.70 (0.063) | 1.76 (0.248) | 1.69 (0.192) | 1.81 (0.209) | 1.99 (0.354) | 1.66 (0.110) | 1.85 (0.214) | 1.85 (0.151) | 1.88 (0.235) | 1.92 (0.210) | 1.95 (0.384) | 1.97 (0.262) | 1.70 (0.250) | 1.72 (0.253) | 1.80 (0.217) | 1.68 (0.154) | 1.82 (0.256) | 1.71 (0.170) | 1.79 (0.219)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of TAK-117
Description: MTD is highest dose level of TAK-117 at which no more than 1 out of 6 participants had a dose limiting toxicity (DLT) during first cycle. DLT was any 1 of following events occurring within first 21 days of Cycle 1 of TAK-117 administration, Grade 2: fasting hyperglycemia for >14 days. Grade 3: nausea and/or vomiting/diarrhea for >7 days; rash for >7 days; thrombocytopenia with bleeding; fasting hyperglycemia for >24 hours(hr). Grade >=3:nonhematologic toxicity considered clinically significant by investigator. Grade 4:neutropenia (absolute neutrophil count <=0.5*10^9per liter[/L]) for >7 days in absence of growth factor support; neutropenia of any duration accompanied with fever >=38.5 degree Celsius and/or systemic infection. Grade >=4:hematologic toxicity. Inability to administer at least 75% of planned doses of TAK-117 within Cycle 1 due to its related toxicity;Any clinically significant occurrence that investigators and sponsor agreed would place participants at undue safety risk.
Time Frame: Baseline up to Cycle 1 Day 21
Population: The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Number; unit: mg
Groups:
- Process A: Total QD TAK-117 100-300 mg: TAK-117 100-300 mg, capsules (Process A), orally, QD up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process A: Total MWF QW 200-1200 mg: TAK-117 200-1200 mg, capsules (Process A), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process A: Total MTW QW 200-900 mg: TAK-117 200-900 mg, capsules (Process A), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days.
- Process B: Total FM MWF QW TAK-117 600-1200 mg: TAK-117 600-1200 mg, capsules (Process B), orally, once every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: Total FM MTW QW 600-1500 mg: TAK-117 600-1500 mg, capsules (Process B), orally, QD for 3 consecutive days, on MTW QW up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
- Process B: Total FM BID MWF QW 300-600 mg: TAK-117 300-600 mg, capsules (Process B), orally, BID every other day on MWF QW up to Day 15 of each treatment cycle. Treatment cycle were repeated every 21 days. FM used drug substance manufactured by an improved synthetic process.
Arm/Group | Process A: Total QD TAK-117 100-300 mg | Process A: Total MWF QW 200-1200 mg | Process A: Total MTW QW 200-900 mg | Process B: Total FM MWF QW TAK-117 600-1200 mg | Process B: Total FM MTW QW 600-1500 mg | Process B: Total FM BID MWF QW 300-600 mg
Number analyzed (Participants) | 24 | 27 | 20 | 13 | 15 | 26
mg | 150 | 900 | 900 | NA — The MTD was not determined because PK data for FM showed limited increase in exposure above 900 mg. | NA — The MTD was not determined because PK data for FM showed limited increase in exposure above 900 mg. | 500

2. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Death, Adverse Events (AEs) Leading to Discontinuation of Study Drug, and DLTs in Cycle 1
Time Frame: Baseline up to Cycle 27 Day 45
Population: The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Number; unit: participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
participants
  TEAE | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 3 | 4 | 10 | 7
  SAE | 2 | 3 | 4 | 2 | 0 | 2 | 0 | 2 | 5 | 2 | 0 | 1 | 0 | 7 | 1 | 2 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 5 | 5
  AEs leading to discontinuation of study drug | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 4
  Death | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  DLTs in Cycle 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Highest Level of TEAEs Severity
Description: Severity of AEs was evaluated based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0 as follow: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (life-threatening); Grade 5 (fatal).
Time Frame: Baseline up to Cycle 27 Day 45
Population: The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Number; unit: participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
participants
  Grade 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 3 | 4 | 2 | 1 | 1 | 2 | 2 | 2 | 5 | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 3 | 3 | 0 | 0 | 3 | 1 | 1 | 4 | 1
  Grade 3 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 5 | 3 | 1 | 1 | 1 | 7 | 1 | 1 | 3 | 0 | 2 | 1 | 3 | 1 | 2 | 3 | 4
  Grade 4 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  Grade 5 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Laboratory Values
Time Frame: Baseline up to Cycle 27 Day 45
Population: The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Number; unit: participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs
Time Frame: Baseline up to Cycle 27 day 45
Population: The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Number; unit: participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Electrocardiogram (ECG)
Time Frame: Baseline up to Cycle 27 Day 45
Population: The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Number; unit: participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Response Rate (ORR)
Description: The estimate of the ORR is calculated as crude percentage of participants who's best overall response is complete response (CR) or partial response (PR). Objective response (CR and PR) as determined by the participants best tumor response was assessed using response evaluation criteria in solid tumors (RECIST) version 1.1. As per RECIST version 1.1, CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 millimeter [mm]). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease was defined as not qualifying for CR, PR, and progressive disease (PD).
Time Frame: Cycle 1 Day 8 up to Cycle 27 Day 1 or disease progression or death
Population: The full analysis set (FAS) population included participants who received at least 1 dose of TAK-117, baseline data for those analyses that required baseline data and postbaseline endpoint data subsequent to at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 4 | 6 | 8 | 2 | 3 | 3 | 3 | 3 | 10 | 3 | 3 | 3 | 1 | 9 | 3 | 1 | 5 | 3 | 2 | 3 | 5 | 3 | 3 | 8 | 4
percentage of participants | 0 [0.00 to 60.24] | 0 [0.00 to 45.93] | 13 [0.32 to 52.65] | 100 [15.81 to 100.00] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 30.85] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 97.50] | 0 [0.00 to 33.63] | 0 [0.00 to 70.76] | 0 [0.00 to 97.50] | 0 [0.00 to 52.18] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 70.76] | 0 [0.00 to 52.18] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 36.94] | 25 [0.63 to 80.59]

8. Secondary Outcome: Duration of Objective Response
Description: Duration of response was to be calculated for participants who achieved CR or PR. Duration of objective response was defined as the number of days from the start date of PR or CR (whichever response was achieved first) to the first date that PD or disease progression was objectively documented. The duration of objective response was to be right-censored for participants who achieved CR or PR and met 1 of the following conditions: Non-protocol anticancer treatment started before documentation of PD; Documented PD after more than 1 missed disease assessment visit; Alive and did not have documentation of PD before a data analysis cutoff date.
Time Frame: Cycle 1 Day 8 up to Cycle 27 Day 1 or disease progression or death
Population: The duration of objective response analysis was not performed due to change in planned analysis.
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate was defined as the participants who achieved stable disease (SD) for at least 15 weeks, CR, or PR. The estimate of the CBR was calculated as crude percentage of participants whose best ORR was CR, PR or SD for at least 90 days.
Time Frame: Cycle 1 Day 8 up to Cycle 27 Day 1 or disease progression or death
Population: The FAS population included participants who received at least 1 dose of TAK-117, baseline data for those analyses that required baseline data and postbaseline endpoint data subsequent to at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 4 | 6 | 8 | 2 | 3 | 3 | 3 | 3 | 10 | 3 | 3 | 3 | 1 | 9 | 3 | 1 | 5 | 3 | 2 | 3 | 5 | 3 | 3 | 8 | 4
percentage of participants | 25 [0.63 to 80.59] | 17 [0.42 to 64.12] | 38 [8.52 to 75.51] | 100 [15.81 to 100.00] | 33 [0.84 to 90.57] | 33 [0.84 to 90.57] | 33 [0.84 to 90.57] | 0 [0.00 to 70.76] | 20 [2.52 to 55.61] | 67 [9.43 to 99.16] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 97.50] | 56 [21.20 to 86.30] | 33 [0.84 to 90.57] | 0 [0.00 to 97.50] | 0 [0.00 to 52.18] | 33 [0.84 to 90.57] | 0 [0.00 to 84.19] | 0 [0.00 to 70.76] | 0 [0.00 to 52.18] | 0 [0.00 to 70.76] | 33 [0.84 to 90.57] | 25 [3.19 to 65.09] | 25 [0.63 to 80.59]

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-117
Time Frame: Process A: Cycle 1 Day 1 pre-dose and at multiple timepoints (up to 24 hrs) post-dose; Process B: Cycle 1 Day 1 pre-dose and at multiple timepoints (up to 48 hrs) post-dose
Population: Pharmacokinetic (PK) population included all participants who took at least 1 dose of study drug and had sufficient plasma concentration-time data to calculate PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Process A: TAK-117 100 mg: Cohort 1: TAK-117 100 mg, capsules, orally, once a day (QD), continuously for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 150 mg: Cohort 2: TAK-117 150 mg, capsules, orally, QD, continuously for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 200 mg: Cohort 3: TAK-117 200 mg, capsules, orally, QD, continuously; Cohort 5: TAK-117 200 mg, capsules, orally, intermittently, once every other day on MWF QW; Cohort 11: TAK-117 200 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW. TAK-117 was administered in all 3 cohorts for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 300 mg: Cohort 4: TAK-117 300 mg, capsules, orally, QD, continuously; Cohort 6: TAK-117 300 mg, capsules, orally, intermittently, once every other day on MWF QW. TAK-117 was administered in both the cohorts for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 400 mg: Cohort 7: TAK-117 400 mg, capsules, orally, intermittently, once every other day on MWF QW; Cohort 12: TAK-117 400 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW. TAK-117 was administered in both the cohorts for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 600 mg: Cohort 8: TAK-117 600 mg, capsules, orally, intermittently, once every other day on MWF QW; Cohort 13: TAK-117 600 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW. TAK-117 was administered in both the cohorts for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 900 mg: Cohort 9: TAK-117 900 mg, capsules, orally, intermittently, once every other day on MWF QW; Cohort 14: TAK-117 200 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW. TAK-117 was administered in both the cohorts for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process A: TAK-117 1200 mg: Cohort 10: TAK-117 1200 mg, capsules, orally, intermittently, once every other day on MWF QW for first 21 days of therapy (Cycle 1). Process A included participants who received original formulation of TAK-117 capsules.
- Process B: TAK-117 300 mg: Cohort 22: TAK-117 300 mg, capsules, orally, intermittently, BID every other day on MWF QW for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 400 mg: Cohort 23: TAK-117 400 mg, capsules, orally, intermittently, BID every other day on MWF QW for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 500 mg: Cohort 24: TAK-117 500 mg, capsules, orally, intermittently, BID every other day on MWF QW for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 600 mg: Cohort 15: TAK-117 600 mg, capsules, orally, intermittently, once every other day on MWF QW; Cohort 18: TAK-117 600 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW; Cohort 25: TAK-117 600 mg, capsules, orally, intermittently, BID every other day on MWF QW. TAK-117 was administered in all the 3 cohorts for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 900 mg: Cohort 16: TAK-117 900 mg, capsules, orally, intermittently, once every other day on MWF QW; Cohort 19: TAK-117 900 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW. TAK-117 was administered in both the cohorts for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 1200 mg: Cohort 17: TAK-117 1200 mg, capsules, orally, intermittently, once every other day on MWF QW ; Cohort 20: TAK-117 1200 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW. TAK-117 was administered in both the cohorts for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
- Process B: TAK-117 1500 mg: Cohort 21: TAK-117 1500 mg, capsules, orally, intermittently, QD for 3 consecutive days, on MTW QW for first 21 days of therapy (Cycle 1). Process B in the study is referred to the study design when new CTM was introduced. FM used drug substance manufactured by an improved synthetic process.
Arm/Group | Process A: TAK-117 100 mg | Process A: TAK-117 150 mg | Process A: TAK-117 200 mg | Process A: TAK-117 300 mg | Process A: TAK-117 400 mg | Process A: TAK-117 600 mg | Process A: TAK-117 900 mg | Process A: TAK-117 1200 mg | Process B: TAK-117 300 mg | Process B: TAK-117 400 mg | Process B: TAK-117 500 mg | Process B: TAK-117 600 mg | Process B: TAK-117 900 mg | Process B: TAK-117 1200 mg | Process B: TAK-117 1500 mg
Number analyzed (Participants) | 6 | 6 | 14 | 7 | 6 | 6 | 23 | 2 | 4 | 4 | 10 | 14 | 6 | 10 | 6
nanogram per milliliter (ng/mL) | 1747.61 (48.7) [0.63 to 80.59] | 1613.23 (58.5) [0.42 to 64.12] | 2736.60 (36.4) [8.52 to 75.51] | 2658.23 (90.0) [15.81 to 100.00] | 4335.88 (42.5) [0.84 to 90.57] | 4175.13 (82.4) [0.84 to 90.57] | 7863.36 (42.1) [0.84 to 90.57] | 8586.50 (53.6) [0.00 to 70.76] | 1162.06 (117.5) [2.52 to 55.61] | 1656.71 (77.0) [9.43 to 99.16] | 2973.26 (53.3) [0.00 to 70.76] | 3870.43 (61.1) [0.00 to 70.76] | 6960.06 (69.3) [0.00 to 97.50] | 6073.55 (53.2) [21.20 to 86.30] | 6899.80 (67.9) [0.84 to 90.57]

11. Secondary Outcome: Ctrough: Observed Concentration at the End of Dosing Interval for TAK-117
Time Frame: as for outcome 10
Population: PK population included all participants who took at least 1 dose of study drug and had sufficient concentration-time data to calculate PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Process A: TAK-117 100 mg | Process A: TAK-117 150 mg | Process A: TAK-117 200 mg | Process A: TAK-117 300 mg | Process A: TAK-117 400 mg | Process A: TAK-117 600 mg | Process A: TAK-117 900 mg | Process A: TAK-117 1200 mg | Process B: TAK-117 300 mg | Process B: TAK-117 400 mg | Process B: TAK-117 500 mg | Process B: TAK-117 600 mg | Process B: TAK-117 900 mg | Process B: TAK-117 1200 mg | Process B: TAK-117 1500 mg
Number analyzed (Participants) | 6 | 6 | 14 | 7 | 6 | 6 | 23 | 2 | 4 | 4 | 10 | 14 | 6 | 10 | 6
ng/mL | 187.29 (102.1) [0.63 to 80.59] | 177.70 (124.0) [0.42 to 64.12] | 630.82 (70.0) [8.52 to 75.51] | 627.62 (93.7) [15.81 to 100.00] | NA (NA) [0.84 to 90.57] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.84 to 90.57] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.84 to 90.57] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.00 to 70.76] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [2.52 to 55.61] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [9.43 to 99.16] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.00 to 70.76] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.00 to 70.76] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.00 to 97.50] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [21.20 to 86.30] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.84 to 90.57] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification.

12. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-117
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Median (Full Range); unit: hr
Arm/Group | Process A: TAK-117 100 mg | Process A: TAK-117 150 mg | Process A: TAK-117 200 mg | Process A: TAK-117 300 mg | Process A: TAK-117 400 mg | Process A: TAK-117 600 mg | Process A: TAK-117 900 mg | Process A: TAK-117 1200 mg | Process B: TAK-117 300 mg | Process B: TAK-117 400 mg | Process B: TAK-117 500 mg | Process B: TAK-117 600 mg | Process B: TAK-117 900 mg | Process B: TAK-117 1200 mg | Process B: TAK-117 1500 mg
Number analyzed (Participants) | 6 | 6 | 14 | 7 | 6 | 6 | 23 | 2 | 4 | 4 | 10 | 14 | 6 | 10 | 6
hr | 1.5 [1 to 4] | 1.5 [1 to 2] | 2.0 [1 to 4] | 2.1 [1 to 4] | 4.0 [1 to 8] | 3.1 [1 to 4] | 2.0 [1 to 8] | 5.8 [4 to 8] | 1.6 [1 to 4] | 4.0 [2 to 8] | 3.6 [2 to 6] | 3.4 [1 to 8] | 4.0 [1 to 8] | 4.0 [1 to 23] | 3.8 [2 to 8]

13. Secondary Outcome: T 1/2z: Terminal Disposition Phase Half-life for TAK-117
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Process A: TAK-117 100 mg | Process A: TAK-117 150 mg | Process A: TAK-117 200 mg | Process A: TAK-117 300 mg | Process A: TAK-117 400 mg | Process A: TAK-117 600 mg | Process A: TAK-117 900 mg | Process A: TAK-117 1200 mg | Process B: TAK-117 300 mg | Process B: TAK-117 400 mg | Process B: TAK-117 500 mg | Process B: TAK-117 600 mg | Process B: TAK-117 900 mg | Process B: TAK-117 1200 mg | Process B: TAK-117 1500 mg
Number analyzed (Participants) | 6 | 6 | 14 | 7 | 6 | 6 | 23 | 2 | 4 | 4 | 10 | 14 | 6 | 10 | 6
hrs | 8.74 (3.0) [0.63 to 80.59] | 7.32 (3.3) [0.42 to 64.12] | 11.17 (4.5) [8.52 to 75.51] | 9.75 (5.5) [15.81 to 100.00] | 12.24 (3.9) [0.84 to 90.57] | 14.71 (6.4) [0.84 to 90.57] | 11.12 (3.9) [0.84 to 90.57] | 25.87 (22.7) [0.00 to 70.76] | NA (NA) [2.52 to 55.61] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [9.43 to 99.16] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.00 to 70.76] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | 12.17 (4.0) [0.00 to 70.76] | 8.34 (4.7) [0.00 to 97.50] | 14.28 (3.5) [21.20 to 86.30] | 9.53 (2.5) [0.84 to 90.57]

14. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-117
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | Process A: TAK-117 100 mg | Process A: TAK-117 150 mg | Process A: TAK-117 200 mg | Process A: TAK-117 300 mg | Process A: TAK-117 400 mg | Process A: TAK-117 600 mg | Process A: TAK-117 900 mg | Process A: TAK-117 1200 mg | Process B: TAK-117 300 mg | Process B: TAK-117 400 mg | Process B: TAK-117 500 mg | Process B: TAK-117 600 mg | Process B: TAK-117 900 mg | Process B: TAK-117 1200 mg | Process B: TAK-117 1500 mg
Number analyzed (Participants) | 6 | 6 | 14 | 7 | 6 | 6 | 23 | 2 | 4 | 4 | 10 | 14 | 6 | 10 | 6
nanogram hours per milliliter (ng*hr/mL) | 18008 (78.8) [0.63 to 80.59] | 13807 (93.2) [0.42 to 64.12] | 44733 (58.0) [8.52 to 75.51] | 42909 (102.2) [15.81 to 100.00] | 93748 (19.8) [0.84 to 90.57] | 75937 (94.4) [0.84 to 90.57] | 129217 (56.0) [0.84 to 90.57] | 309073 (23.7) [0.00 to 70.76] | NA (NA) [2.52 to 55.61] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [9.43 to 99.16] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | NA (NA) [0.00 to 70.76] — Values were not estimable since serum concentration of TAK-117 were below the limit of quantification. | 62876 (78.4) [0.00 to 70.76] | 84394 (103.1) [0.00 to 97.50] | 164508 (74.9) [21.20 to 86.30] | 87515 (81.2) [0.84 to 90.57]

15. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-117
Time Frame: as for outcome 10
Population: No data is reported since serum concentration of TAK-117 were below the limit of quantification.
Arm/Group | Process A: TAK-117 100 mg | Process A: TAK-117 150 mg | Process A: TAK-117 200 mg | Process A: TAK-117 300 mg | Process A: TAK-117 400 mg | Process A: TAK-117 600 mg | Process A: TAK-117 900 mg | Process A: TAK-117 1200 mg | Process B: TAK-117 300 mg | Process B: TAK-117 400 mg | Process B: TAK-117 500 mg | Process B: TAK-117 600 mg | Process B: TAK-117 900 mg | Process B: TAK-117 1200 mg | Process B: TAK-117 1500 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: %AUC Extrapolated: Percentage of Area Under Concentration-extrapolated
Time Frame: as for outcome 10
Population: No data is reported since serum concentration of TAK-117 were below the limit of quantification.
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Percent Change From Baseline in Pharmacodynamic Markers
Description: Pharmacodynamic markers included phosphorylated ribosomal protein S6 (PS6), phosphorylated eukaryotic initiation factor 4E-binding protein 1 (P4EBP1), phosphorylated N-myc downstream regulated gene 1 (PNDRG1), phosphorylated proline-rich AKT substrate of 40 kilodaltons (PPRAS40), and phosphorylated serine/threonine protein kinase AKT (PAKT). Analysis population (n) for each skin biopsy biomarker is as follow: P4EBP1 (n=6,6,6,2,2,0,0,0,0,1,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0); PAKT and PNDRG1 (n=6,6,7,2,2,0,0,0,0,1,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0); PPRAS40 (n= 6,0,6,2,2,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0); PS6 (n=6,6,7,2,2,0,0,0,0,1,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0)."n" for each tumor tissue biomarkers is as follow: P4EBP1, PAKT, PNDRG1, and PS6 (n=1,1,0,0,1,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0); PPRAS40 (n= 1,0,0,0,1,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0,0).
Time Frame: Cycle 1 Day 8
Population: Asat population where baseline and post-baseline assessments were available. The ASat population included all enrolled participants who received at least 1 dose of TAK-117.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 3 | 3 | 3 | 3 | 12 | 3 | 3 | 3 | 3 | 11 | 3 | 3 | 7 | 3 | 3 | 3 | 6 | 4 | 4 | 10 | 8
percent change
  Skin Biopsy: P4EBP1 | -27.94 (56.666) | -13.07 (39.758) | -61.41 (40.015) | -24.50 (54.388) | -100.00 (0.000) | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | -100.00 (NA) — Standard deviation could not be calculate since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category.
  Skin Biopsy: PAKT | -11.59 (33.833) | 190.32 (257.212) | -30.02 (37.444) | -12.97 (5.896) | -18.75 (26.517) | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | 733.33 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category.
  Skin Biopsy: PNDRG1 | -9.82 (15.138) | -0.11 (35.915) | -10.11 (26.814) | -21.67 (35.355) | 10.69 (31.283) | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | -34.44 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category.
  Skin Biopsy: PPRAS40 | 69.56 (272.327) | NA (NA) — None of the participants were evaluable for this category. | -26.90 (37.191) | -18.75 (61.872) | -14.17 (8.250) | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category. | NA (NA) — None of the participants were evaluable for this category.
  Skin Biopsy: PS6 | -15.23 (18.886) | -25.05 (15.883) | -11.88 (37.773) | 22.70 (24.462) | 9.54 (19.146) | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | 46.15 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis.
  Tumor Tissue: P4EBP1 | 236.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | -97.56 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | 7.48 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis.
  Tumor Tissue: PAKT | 850.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | -20.87 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | -44.83 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis.
  Tumor Tissue: PNDRG1 | 134.69 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | -16.49 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | 134.29 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis.
  Tumor Tissue: PPRAS40 | 196.83 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | 10.43 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis.
  Tumor Tissue: PS6 | 200.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.00 (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | -82.86 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis. | NA (NA) — Data was not calculated since no participant was available for analysis.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) | Process A: TAK-117 150 mg, QD | Process A: TAK-117 200 mg, QD | Process A: TAK-117 300 mg, QD | Process A: TAK-117 200 mg, MWF QW | Process A: TAK-117 300 mg, MWF QW | Process A: TAK-117 400 mg, MWF QW | Process A: TAK-117 600 mg, MWF QW | Process A: TAK-117 900 mg, MWF QW | Process A: TAK-117 1200 mg, MWF QW | Process A: TAK-117 200 mg, MTW QW | Process A: TAK-117 400 mg, MTW QW | Process A: TAK-117 600 mg, MTW QW | Process A: TAK-117 900 mg, MTW QW | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW | Process B: TAK-117 900 mg FM MWF QW | Process B: TAK-117 1200 mg FM MWF QW | Process B: TAK-117 600 mg FM MTW QW | Process B: TAK-117 900 mg FM MTW QW | Process B: TAK-117 1200 mg FM MTW QW | Process B: TAK-117 1500 mg FM MTW QW | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW | Process B: TAK-117 400 mg FM BID MWF QW | Process B: TAK-117 500 mg FM BID MWF QW | Process B: TAK-117 600 mg FM BID MWF QW
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 4/8 | 2/4 | 0/3 | 2/3 | 0/3 | 2/3 | 5/12 | 2/3 | 0/3 | 1/3 | 0/3 | 7/11 | 1/3 | 2/3 | 2/7 | 1/3 | 1/3 | 1/3 | 2/6 | 1/4 | 1/4 | 5/10 | 5/8
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 8/8 | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 12/12 | 3/3 | 3/3 | 3/3 | 3/3 | 11/11 | 3/3 | 3/3 | 7/7 | 3/3 | 3/3 | 3/3 | 6/6 | 2/4 | 4/4 | 10/10 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) (N=6) | Process A: TAK-117 150 mg, QD (N=6) | Process A: TAK-117 200 mg, QD (N=8) | Process A: TAK-117 300 mg, QD (N=4) | Process A: TAK-117 200 mg, MWF QW (N=3) | Process A: TAK-117 300 mg, MWF QW (N=3) | Process A: TAK-117 400 mg, MWF QW (N=3) | Process A: TAK-117 600 mg, MWF QW (N=3) | Process A: TAK-117 900 mg, MWF QW (N=12) | Process A: TAK-117 1200 mg, MWF QW (N=3) | Process A: TAK-117 200 mg, MTW QW (N=3) | Process A: TAK-117 400 mg, MTW QW (N=3) | Process A: TAK-117 600 mg, MTW QW (N=3) | Process A: TAK-117 900 mg, MTW QW (N=11) | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW (N=3) | Process B: TAK-117 900 mg FM MWF QW (N=3) | Process B: TAK-117 1200 mg FM MWF QW (N=7) | Process B: TAK-117 600 mg FM MTW QW (N=3) | Process B: TAK-117 900 mg FM MTW QW (N=3) | Process B: TAK-117 1200 mg FM MTW QW (N=3) | Process B: TAK-117 1500 mg FM MTW QW (N=6) | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW (N=4) | Process B: TAK-117 400 mg FM BID MWF QW (N=4) | Process B: TAK-117 500 mg FM BID MWF QW (N=10) | Process B: TAK-117 600 mg FM BID MWF QW (N=8)
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Process A: TAK-117 100 Milligram (mg), Once Daily (QD) (N=6) | Process A: TAK-117 150 mg, QD (N=6) | Process A: TAK-117 200 mg, QD (N=8) | Process A: TAK-117 300 mg, QD (N=4) | Process A: TAK-117 200 mg, MWF QW (N=3) | Process A: TAK-117 300 mg, MWF QW (N=3) | Process A: TAK-117 400 mg, MWF QW (N=3) | Process A: TAK-117 600 mg, MWF QW (N=3) | Process A: TAK-117 900 mg, MWF QW (N=12) | Process A: TAK-117 1200 mg, MWF QW (N=3) | Process A: TAK-117 200 mg, MTW QW (N=3) | Process A: TAK-117 400 mg, MTW QW (N=3) | Process A: TAK-117 600 mg, MTW QW (N=3) | Process A: TAK-117 900 mg, MTW QW (N=11) | Process B: TAK-117 600 mg Process B Capsule (FM) MWF QW (N=3) | Process B: TAK-117 900 mg FM MWF QW (N=3) | Process B: TAK-117 1200 mg FM MWF QW (N=7) | Process B: TAK-117 600 mg FM MTW QW (N=3) | Process B: TAK-117 900 mg FM MTW QW (N=3) | Process B: TAK-117 1200 mg FM MTW QW (N=3) | Process B: TAK-117 1500 mg FM MTW QW (N=6) | Process B: TAK-117 300 mg FM Twice Daily (BID) MWF QW (N=4) | Process B: TAK-117 400 mg FM BID MWF QW (N=4) | Process B: TAK-117 500 mg FM BID MWF QW (N=10) | Process B: TAK-117 600 mg FM BID MWF QW (N=8)
Nausea (Gastrointestinal disorders) | 3 | 4 | 5 | 2 | 1 | 2 | 0 | 3 | 8 | 1 | 2 | 2 | 1 | 10 | 2 | 1 | 6 | 1 | 2 | 2 | 4 | 2 | 2 | 7 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 2 | 2 | 0 | 2 | 8 | 2 | 2 | 1 | 2 | 7 | 0 | 2 | 5 | 1 | 2 | 0 | 4 | 2 | 1 | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 5 | 3 | 0 | 1 | 2 | 1 | 6 | 1 | 0 | 0 | 2 | 8 | 0 | 2 | 5 | 0 | 1 | 1 | 4 | 2 | 2 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 4 | 3 | 1 | 1 | 0 | 1 | 2 | 4 | 1 | 1 | 1 | 0 | 4 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4 | 2 | 1 | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 4 | 0 | 1 | 4 | 1 | 0 | 1 | 3 | 1 | 3 | 6 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 4 | 2 | 1 | 1 | 1 | 6 | 2 | 0 | 2 | 1 | 1 | 0 | 3 | 1 | 2 | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 6 | 4 | 1 | 1 | 2 | 1 | 0 | 7 | 1 | 3 | 1 | 0 | 6 | 0 | 2 | 3 | 2 | 2 | 3 | 5 | 1 | 1 | 6 | 2
Asthenia (General disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 4 | 3 | 2 | 2 | 1 | 0 | 4 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 3
Alanine aminotransferase increased (Investigations) | 1 | 2 | 3 | 3 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 4
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insulin C-peptide decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric pH decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting psychogenic (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Portal vein occlusion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.